CLINICAL TRIAL: NCT00660556
Title: Compassionate Use Supplement to the IDE Protocol to Determine Safety and Effectiveness of the ARCHIMEDES Implantable Constant-Flow Infusion Pump System
Brief Title: ARCHIMEDES Compassionate Use Supplement
Status: No longer available | Type: Expanded Access
Sponsor: Cerenovus, Part of DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DDS-US02-001
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Pain
Keywords: Implantable pump; Intrathecal catheter; Constant flow pump
MeSH Terms: conditions — Pain | interventions — Drug Delivery Systems

INTERVENTIONS:
Device: Archimedes Constant Flow Pump & System — Pump implanted in abdomen with intrathecal delivery (catheter) for pain.

SUMMARY:
The purpose of this Compassionate Use Supplement to the IDE Protocol is to assure and monitor the safety of six Subjects (in the United States) implanted with ARCHIMEDES until all remaining implanted pumps are explanted.

DETAILED DESCRIPTION:
Pain management has been a long-standing challenge to the medical community, specifically the treatment of chronic pain. On October 3, 2002, FDA approved Codman's IDE Study of Codman's Implantable Constant-Flow Infusion Pump System (ARCHIMEDES). The first Subject was implanted on February 12, 2003. Since then, ten Subjects have had the ARCHIMEDES implanted, with one Subject, implanted twice. Codman notified the FDA in 2004 that it wished to discontinue enrollment into the study & bring it to a close because of projected slow enrollment and waning physician interest.

Codman felt there was no readily acceptable alternate therapy that would not require a pump explant first. It is possible to replace the ARCHIMEDES with another pump system, which is already approved for use in the United States. However, such an action would necessitate the removal or explant of the ARCHIMEDES, thereby exposing the Subjects to additional risks inherent in such a surgical procedure, including those associated with anesthesia. Since these Subjects have been treated with the investigational device for at least 2 years without experiencing any unanticipated adverse device effects, Codman felt that the risk of explanting the pump was significantly greater than the risk of continuing treatment with the investigational device.

It should also be noted that this pump does not have a battery and that replacement is dictated by the number of times the septum is punctured (500). This translates into approximately twenty years of therapy if the septum is punctured an average of 20 times.

FDA approved Codman's Compassionate Use Protocol in 2005.

ELIGIBILITY:
Inclusion Criteria:

* U. S. Subjects implanted with constant flow pump in 2003.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- South Side Pain Solutions, Danville, Virginia, United States